CLINICAL TRIAL: NCT03005379
Title: CSP #2004 - Microbiota or Placebo After Antimicrobial Therapy for Recurrent C. Difficile at Home (MATCH)
Brief Title: Microbiota or Placebo After Antimicrobial Therapy for Recurrent C. Difficile at Home (MATCH)
Acronym: MATCH
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study is terminated for futility per protocol-specified interim analysis and DMC recommendation.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2004
Record Dates: First submitted 2016-12-14; First posted 2016-12-29 (Estimated); Results first posted 2023-10-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-03

CONDITIONS: Clostridium Difficile Infection
Keywords: FMT; recurrent c. difficile; infectious disease; intestine; clinical trial; gastrointestinal; prevention; randomized; diarrhea; fecal microbiota therapy
MeSH Terms: conditions — Clostridium Infections; Communicable Diseases; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 (Active Comparator): Fecal Microbiota Therapy (FMT)
  Interventions: Drug: Fecal Microbiota Therapy (FMT)
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fecal Microbiota Therapy (FMT) — Oral capsule-delivered FMT
  Arms: 1
Drug: Placebo — Oral capsule-delivered placebo
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether Fecal Microbiota Therapy (FMT) is effective vs. placebo in the prevention of C. difficile infection recurrence.

DETAILED DESCRIPTION:
Clostridium difficile infection (CDI) is one of the most common nosocomial infections and is increasingly seen in non-hospitalized patients. Although more than 90% of patients have symptom resolution with a course of standard antimicrobial therapy, subsequent recurrence rates range from 15-30% (after the first CDI episode) to 40-50% (after the second and subsequent episodes). Fecal microbiota transplantation (FMT) has shown promise as an adjunct to standard antimicrobial therapy, reducing recurrence among FMT recipients to 15%.

The primary study goal is to assess the efficacy of FMT for the prevention of subsequent recurrent CDI, when administered after successful treatment of recurrent CDI with standard antimicrobial therapy. Secondary goals are to evaluate, the efficacy of FMT in terms of CDI severity, duration, the safety of FMT, and in the event of a positive study result, establish a mechanism for providing FMT within the VA system.

This study will enroll 390 participants. Participants will be randomized (1:1 ratio) to FMT or placebo, stratified by number of prior recurrent CDI episodes (1 versus >1). They will be assessed for symptoms of CDI, other study outcomes and any treatment-related adverse events at 2, 14, 28, 42, and 56 days, and month 3, 4, 5 and 6 after administration of the study treatment.

The primary outcome is recurrent CDI (definite or possible) or death within 56 days of randomization.

Definite recurrence is defined as any of the following: The new onset of more than three loose or watery stools in 24 hours for two consecutive days, not explained by another diagnosis; Other clinical symptoms including ileus, toxic megacolon, or colectomy; plus laboratory confirmation of C. difficile from a stool specimen by toxin Enzyme Immunoassays (EIA) test. Possible recurrence is defined as the same clinical manifestations as above, but without laboratory confirmation of C. difficile (stool test not sent, negative EIA toxin test result, or uninterpretable result).

ELIGIBILITY:
Inclusion Criteria:

1. One or more episodes recurrent CDI (defined as > 3 loose/watery stools/24h for 2 consecutive days with CDI treatment, and not explained by another diagnosis plus laboratory confirmation of C. difficile; or ileus, or toxic megacolon plus laboratory confirmation of C. difficile, occurring within 90 days of a prior CDI episode with similar symptoms and laboratory confirmation)
2. Resolution or improvement of symptoms from most recent CDI episode, defined as no longer meeting the clinical definition for CDI for a 48 hour period during treatment, including not meeting the definition again after an initial improvement
3. Within the enrollment window: 2 days after completion of antimicrobial therapy for CDI (to allow for a washout period) to 14 days after completion of therapy or 30 days after the onset of CDI whichever is later.
4. Age 18 years
5. Enrolled in a Veterans Health Administration (VHA) facility
6. Able and willing to provide informed consent

Exclusion Criteria:

1. Unlikely to swallow capsules
2. Pregnancy, planning to be pregnant, or breastfeeding
3. Receipt of cytotoxic chemotherapy, intravenous or subcutaneous immune globulin, or confirmed neutropenia (absolute neutrophil count of < 1,000 cells/ L) within the past 3 months
4. Inflammatory bowel disease or other chronic diarrheal disease/fecal incontinence predating CDI
5. Ongoing antibiotic use other than those for the current episode of CDI
6. Prior FMT
7. Life expectancy of < 8 weeks
8. Anaphylactic food allergy
9. Active enrollment in another research study on antibiotics, probiotics, or FMT without investigators approval
10. Presence of an ileostomy or colostomy
11. HIV with Clusters of Differentiation 4 (CD4) cell count < 200 cells/µL in prior 3 months
12. Decompensated cirrhosis
13. Bone marrow/peripheral blood stem cell transplant in the past year
14. Unlikely to follow study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri M Drekonja, MD, Study Chair — Minneapolis VA Health Care System, Minneapolis, MN; Aasma Shaukat, MD MPH, Study Chair — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Digital data underlying primary scientific publications from this study will be held as part of a data sharing resource maintained by the Cooperative Studies Program (CSP). Study data held for this purpose may include data, data content, format, and organization. The data may be available to the public and other VA and non-VA researchers under certain conditions and consistent with the informed consent and CSP policy which prioritize protecting subjects' privacy and confidentiality to the fullest extent possible.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Result] Drekonja DM, Shaukat A, Zhang JH, Reinink AR, Nugent S, Dominitz JA, Davis-Karim A, Gerding DN, Kyriakides TC. Microbiota or placebo after antimicrobial therapy for recurrent Clostridioides difficile at home: A clinical trial with novel home-based enrollment. Clin Trials. 2021 Oct;18(5):622-629. doi: 10.1177/17407745211021198. Epub 2021 Jun 22. PMID 34154439
- [Derived] Drekonja DM, Shaukat A, Huang Y, Zhang JH, Reinink AR, Nugent S, Dominitz JA, Davis-Karim A, Gerding DN, Kyriakides TC. A Randomized Controlled Trial of Efficacy and Safety of Fecal Microbiota Transplant for Preventing Recurrent Clostridioides difficile Infection. Clin Infect Dis. 2025 Feb 5;80(1):52-60. doi: 10.1093/cid/ciae467. PMID 39271107

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study did not contain pre-assignment.
Groups:
- Fecal Microbiota Therapy: Fecal Microbiota Therapy (FMT)
  Fecal Microbiota Therapy (FMT): Oral capsule-delivered FMT
- Placebo: Placebo
  Placebo: Oral capsule-delivered placebo
Period: Overall Study
Arm/Group | Fecal Microbiota Therapy | Placebo
Started | 76 | 77
Completed | 76 | 76
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: all participants who were randomized
Groups:
- Fecal Microbiota Therapy (FMT): Fecal Microbiota Therapy (FMT)
  Fecal Microbiota Therapy (FMT): Oral capsule-delivered FMT
- Total: Total of all reporting groups
Arm/Group | Fecal Microbiota Therapy (FMT) | Placebo | Total
Number analyzed (Participants) | 76 | 77 | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 33 | 53
  >=65 years | 56 | 44 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (12.31) | 63.9 (14.63) | 66.5 (13.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 68 | 64 | 132
Race/Ethnicity, Customized [Number; unit: participants] — Race is a multiple-choice question
  participants
    Race : White | 70 | 75 | 145
    Race : African-American or Black | 6 | 2 | 8
    Race : American Indian or Alaska Native | 3 | 0 | 3
    Race : Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Race : Chinese | 0 | 0 | 0
    Race : Japanese | 0 | 0 | 0
    Race : Filipino | 0 | 0 | 0
    Race : Asian Indian | 0 | 0 | 0
    Race : Other Asian | 0 | 0 | 0
    Race : Other Race | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 76 | 77 | 153
Albumin [Mean (Standard Deviation); unit: g/dL] — Population: baseline labs were not available for a few participants
  g/dL
    number analyzed (Participants) | 71 | 71 | 142
    (all) | 3.7 (0.6) | 3.9 (0.6) | 3.8 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Possible or Definite Recurrent Clostridium Difficile Infection (CDI), or Death
Description: The primary outcome is recurrent CDI (definite or possible) or death within 56 days of randomization.
  A possible CDI recurrence is defined as a new onset of more than three loose or watery stools in 24 hours for two consecutive days, not explained by another diagnosis, other clinical symptoms including ileus, toxic megacolon, or colectomy. As part of the protocol procedures, a possible CDI recurrence is adjudicated by the study's adjudication committee. A definite CDI recurrence is defined as a potential CDI recurrence with symptom (more than three loose or watery stools in 24 hours for two consecutive days, not explained by another diagnosis, other clinical symptoms including ileus, toxic megacolon, or colectomy) plus laboratory confirmation of C. difficile from a stool specimen by toxin Enzyme Immunoassays (EIA) test.
Time Frame: Within 56 days of randomization
Population: All randomized participants are analyzed according to the principle of intent-to-treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota Therapy (FMT) | Placebo
Number analyzed (Participants) | 76 | 77
Participants | 25 | 23

2. Secondary Outcome: Recurrent CDI (Definite or Possible) or Death Within 6 Months of Randomization.
Description: A possible CDI recurrence is defined as a new onset of more than three loose or watery stools in 24 hours for two consecutive days, not explained by another diagnosis, other clinical symptoms including ileus, toxic megacolon, or colectomy. As part of the protocol procedures, a possible CDI recurrence is adjudicated by the study's adjudication committee. A definite CDI recurrence is defined as a potential CDI recurrence with symptom (more than three loose or watery stools in 24 hours for two consecutive days, not explained by another diagnosis, other clinical symptoms including ileus, toxic megacolon, or colectomy) plus laboratory confirmation of C. difficile from a stool specimen by EIA toxin test.
Time Frame: Within 6 months of randomization
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota Therapy (FMT) | Placebo
Number analyzed (Participants) | 76 | 77
Participants | 32 | 31

3. Secondary Outcome: Quality of Life at 56 Day
Description: The investigators will use a brief assessment of both overall and gastrointestinal health status, a previously validated instrument called Gastrointestinal Quality of Life Index (GIQLI). GIQLI takes value between 0 and 144, with higher score associated with better quality of life.
Time Frame: 56 days from randomization
Population: Intent-to-treat & complete-case
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fecal Microbiota Therapy (FMT) | Placebo
Number analyzed (Participants) | 72 | 69
units on a scale | 111.42 (21.25) | 115.67 (19.15)

4. Secondary Outcome: Frequency of Possible CDI Recurrences Within 6 Months of Randomization
Description: A possible CDI recurrence is defined as a new onset of more than three loose or watery stools in 24 hours for two consecutive days, not explained by another diagnosis, other clinical symptoms including ileus, toxic megacolon, or colectomy. As part of the protocol procedures, a possible CDI recurrence is adjudicated by the study's adjudication committee.
Time Frame: Within 6 months of randomization
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota Therapy (FMT) | Placebo
Number analyzed (Participants) | 76 | 77
Participants
  Have no possible CDI recurrence | 45 | 48
  Have one possible CDI recurrence | 23 | 19
  Have two possible CDI recurrences | 7 | 9
  Have three possible CDI recurrences | 1 | 1

5. Secondary Outcome: Diarrhea That is Negative for C. Difficile by EIA Toxin Test and Polymerase Chain Reaction (PCR)
Description: This is similar to a possible recurrent CDI, but includes only episodes of diarrhea that are tested negative for C. difficile by EIA toxin test and PCR. A possible CDI recurrence is defined as a new onset of more than three loose or watery stools in 24 hours for two consecutive days, not explained by another diagnosis, other clinical symptoms including ileus, toxic megacolon, or colectomy. As part of the protocol procedures, a possible CDI recurrence is adjudicated by the study's adjudication committee.
Time Frame: Within 56 days of randomization
Population: intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota Therapy | Placebo
Number analyzed (Participants) | 76 | 77
Participants | 9 | 8

6. Secondary Outcome: Occurrence of Abdominal Pain Among All Possible CDI Recurrences.
Description: A possible CDI recurrence is defined as a new onset of more than three loose or watery stools in 24 hours for two consecutive days, not explained by another diagnosis, other clinical symptoms including ileus, toxic megacolon, or colectomy. As part of the protocol procedures, a possible CDI recurrence is adjudicated by the study's adjudication committee. Participants were asked to report whether they experienced abdominal pain in each of their possible CDI recurrences.
Time Frame: Within 6 months of randomization
Population: intent-to-treat
Measure: Count of Units; unit: Recurrences
Units Other Than Participants: Recurrences
Groups:
- Fecal Microbiota Therapy: All possible CDI recurrences for Fecal Microbiota Therapy (FMT): Oral capsule-delivered FMT
- Placebo: All possible CDI recurrences for Placebo: Oral capsule-delivered placebo
Arm/Group | Fecal Microbiota Therapy | Placebo
Number analyzed (Participants) | 76 | 77
Number analyzed (Recurrences) | 40 | 40
Recurrences | 19 | 24

7. Secondary Outcome: Definite Recurrent CDI
Description: The occurrence of definite recurrent CDI within 56 days of randomization. A definite CDI recurrence is defined as a potential CDI recurrence with symptom (more than three loose or watery stools in 24 hours for two consecutive days, not explained by another diagnosis, other clinical symptoms including ileus, toxic megacolon, or colectomy) plus laboratory confirmation of C. difficile from a stool specimen by EIA toxin test.
Time Frame: Within 56 days of randomization
Population: intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota Therapy | Placebo
Number analyzed (Participants) | 76 | 77
Participants | 6 | 7

8. Secondary Outcome: Possible Recurrent CDI
Description: The occurrence of possible recurrent CDI within 56 days of randomization. A possible CDI recurrence is defined as a new onset of more than three loose or watery stools in 24 hours for two consecutive days, not explained by another diagnosis, other clinical symptoms including ileus, toxic megacolon, or colectomy. As part of the protocol procedures, a possible CDI recurrence is adjudicated by the study's adjudication committee.
Time Frame: Within 56 days of randomization
Population: intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota Therapy | Placebo
Number analyzed (Participants) | 76 | 77
Participants | 24 | 22

9. Secondary Outcome: Death
Description: The occurrence of death within 56 days of randomization.
Time Frame: Within 56 days of randomization
Population: intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota Therapy | Placebo
Number analyzed (Participants) | 76 | 77
Participants | 1 | 1

10. Secondary Outcome: Diarrhea That is Negative for C. Difficile by EIA Toxin Testing But Positive by PCR
Description: This is similar to possible recurrent CDI, but includes only episodes of diarrhea that are tested negative for C. difficile by EIA toxin test but positive by PCR. A possible CDI recurrence is defined as a new onset of more than three loose or watery stools in 24 hours for two consecutive days, not explained by another diagnosis, other clinical symptoms including ileus, toxic megacolon, or colectomy. As part of the protocol procedures, a possible CDI recurrence is adjudicated by the study's adjudication committee.
Time Frame: Within 56 days of randomization
Population: intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota Therapy (FMT) | Placebo
Number analyzed (Participants) | 76 | 77
Participants | 6 | 6

11. Secondary Outcome: Occurrence of Urgency Among All Possible CDI Recurrences.
Description: A possible CDI recurrence is defined as a new onset of more than three loose or watery stools in 24 hours for two consecutive days, not explained by another diagnosis, other clinical symptoms including ileus, toxic megacolon, or colectomy. As part of the protocol procedures, a possible CDI recurrence is adjudicated by the study's adjudication committee. Participants were asked to report whether they experienced urgency in each of their possible CDI recurrences. The urgency is defined as the urgent need to pass stool, feelings of incomplete bowel control, or inability to control defecation.
Time Frame: within 6 months from randomization
Population: intent-to-treat
Measure: Count of Units; unit: Recurrences
Units Other Than Participants: Recurrences
Arm/Group | Fecal Microbiota Therapy | Placebo
Number analyzed (Participants) | 76 | 77
Number analyzed (Recurrences) | 40 | 40
Recurrences | 36 | 36

12. Secondary Outcome: Occurrence of Fecal Incontinence Among All Possible CDI Recurrences.
Description: A possible CDI recurrence is defined as a new onset of more than three loose or watery stools in 24 hours for two consecutive days, not explained by another diagnosis, other clinical symptoms including ileus, toxic megacolon, or colectomy. As part of the protocol procedures, a possible CDI recurrence is adjudicated by the study's adjudication committee. Participants were asked to report whether they experienced fecal incontinence in each of their possible CDI recurrences. Fecal incontinence is defined as having unintentional passing of stool (liquid or solid).
Time Frame: within 6 months from randomization
Population: intent-to-treat
Measure: Count of Units; unit: Recurrences
Units Other Than Participants: Recurrences
Arm/Group | Fecal Microbiota Therapy | Placebo
Number analyzed (Participants) | 76 | 77
Number analyzed (Recurrences) | 40 | 40
Recurrences | 21 | 18

13. Secondary Outcome: Occurrence of Altering Life Style Among All Possible CDI Recurrences
Description: A possible CDI recurrence is defined as a new onset of more than three loose or watery stools in 24 hours for two consecutive days, not explained by another diagnosis, other clinical symptoms including ileus, toxic megacolon, or colectomy. As part of the protocol procedures, a possible CDI recurrence is adjudicated by the study's adjudication committee. Participants were asked to report whether they had to alter their life style (such as using pads) in each of the possible CDI recurrence.
Time Frame: within 6 months of randomization
Population: intent-to-treat
Measure: Count of Units; unit: Recurrences
Units Other Than Participants: Recurrences
Arm/Group | Fecal Microbiota Therapy | Placebo
Number analyzed (Participants) | 76 | 77
Number analyzed (Recurrences) | 40 | 40
Recurrences | 30 | 25

ADVERSE EVENTS:
Time Frame: All participants will be monitored for adverse events from the time of randomization/ administration of study medication to the study exit time (typically at 6 months after study treatment).
Description: The study definition is consistent with those definitions in ClinicalTrials.gov
Arm/Group | Fecal Microbiota Therapy (FMT) | Placebo
All-Cause Mortality (participants affected / at risk) | 1/76 | 5/77
Serious Adverse Events (participants affected / at risk) | 17/76 | 21/77
Other Adverse Events (participants affected / at risk) | 19/76 | 28/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fecal Microbiota Therapy (FMT) (N=76) | Placebo (N=77)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
cardiac failure (Cardiac disorders) | 3 (4) | 1 (1)
atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
faecalomna (Gastrointestinal disorders) | 0 (0) | 1 (1)
haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
vomitting (Gastrointestinal disorders) | 0 (0) | 1 (1)
stent-graft endoleak (General disorders) | 0 (0) | 1 (1)
colicholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
cirrhosis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
solid organ transplant rejection (Immune system disorders) | 1 (1) | 0 (0)
clostridium difficile infection (Infections and infestations) | 2 (2) | 6 (6)
sepsis (Infections and infestations) | 2 (2) | 1 (1)
urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
cellulitis (Infections and infestations) | 2 (2) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
meningitis viral (Infections and infestations) | 0 (0) | 1 (1)
peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
urosepsis (Infections and infestations) | 0 (0) | 1 (1)
colonoscopy (Investigations) | 0 (0) | 1 (1)
metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
major depression (Psychiatric disorders) | 0 (0) | 1 (1)
nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (2)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
peripheral vein occlusion (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fecal Microbiota Therapy (FMT) (N=76) | Placebo (N=77)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (4)
Dafaecation urgency (Gastrointestinal disorders) | 3 (3) | 4 (4)
Flatulence (Gastrointestinal disorders) | 1 (1) | 5 (6)
constipation (Gastrointestinal disorders) | 3 (3) | 3 (3)
diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (3)
abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
abdominal distension (Gastrointestinal disorders) | 0 (0) | 3 (3)
gastrointestinal hypermotility (Gastrointestinal disorders) | 1 (1) | 1 (1)
anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
fatigua (General disorders) | 2 (2) | 0 (0)
pyrexia (General disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
gastritis viral (Infections and infestations) | 0 (0) | 1 (1)
gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
nasopharygnigitis (Infections and infestations) | 0 (0) | 1 (1)
tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
renal function test abnormal (Investigations) | 1 (1) | 0 (0)
white blood cell count increased (Investigations) | 1 (1) | 0 (0)
stool analysis abnormal (Investigations) | 0 (0) | 1 (1)
urine output increased (Investigations) | 0 (0) | 1 (1)
decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 1 (1)
taste disorder (Nervous system disorders) | 0 (0) | 1 (1)
haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/79/NCT03005379/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/79/NCT03005379/SAP_001.pdf
  • Informed Consent Form (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/79/NCT03005379/ICF_002.pdf